CLINICAL TRIAL: NCT06099197
Title: I-CARE 2 RCT: Mobile Telehealth to Reduce Alzheimer'S-related Symptoms for Hispanic Caregivers and Patients
Brief Title: I-CARE 2: Mobile Telehealth to Reduce Alzheimer'S-related Symptoms in Hispanic Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Miriam J Rodriguez, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20311; R01AG078234 (NIH)
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Caregiver Burden; Alzheimer Disease
Keywords: Alzheimer's disease and related dementias; Hispanic caregivers; Caregiver Burden; Behavioral and psychological symptoms of dementia
MeSH Terms: conditions — Caregiver Burden; Alzheimer Disease; Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the Brain CareNotes app or an attention control app.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigator and outcome assessor will be masked to the app assignment (Brain CareNotes vs Attention Control App).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain CareNotes (Experimental): The Brain CareNotes mobile telehealth app is used by unpaid caregivers for BPSD management. It includes remote communication with an external human support person-a care coach-as well as features for users to independently perform health-related activities.
  Interventions: Behavioral: Brain CareNotes
- Attention Control App (Active Comparator): Dementia Guide Expert provides education only and no interactive BPSD management support, coaching, assessment, or external response. It contains "evidence-based expert information on what dementia is, types, contributing factors, risks, symptoms, stages, diagnosis, tests, treatment, management, communication techniques, and links to resources and support services."
  Interventions: Behavioral: Dementia Guide Expert

INTERVENTIONS:
Behavioral: Brain CareNotes — The Brain CareNotes mobile telehealth app is used by unpaid caregivers for BPSD management. It includes remote communication with an external human support person-a care coach-as well as features for users to independently perform health-related activities.
  Arms: Brain CareNotes
Behavioral: Dementia Guide Expert — Dementia Guide Expert provides education only and no interactive BPSD management support, coaching, assessment, or external response. It contains "evidence-based expert information on what dementia is, types, contributing factors, risks, symptoms, stages, diagnosis, tests, treatment, management, communication techniques, and links to resources and support services."
  Arms: Attention Control App

SUMMARY:
This study is a randomized, controlled trial (RCT) to evaluate usability and acceptability, and met and unmet needs from a caregiver intervention app, Brain CareNotes, among unpaid Hispanic caregivers of patients with dementia. Brain CareNotes provides support for management of the behavioral and psychological symptoms of dementia (BPSD) displayed by care recipients. Over 10 months, the trial will enroll 40 Hispanic caregivers of community-dwelling patients diagnosed with Alzheimer's disease or a related dementia (ADRD). Caregivers will be randomized to use the Brain CareNotes app or an attention control education-only app for 12 months, with usage reminders.

DETAILED DESCRIPTION:
This study is a hybrid efficacy-effectiveness RCT to evaluate usability and acceptability, and met and unmet needs from a caregiver intervention app, Brain CareNotes. Over 10 months, the trial will enroll 40 Hispanic caregivers. Participants will be randomized to use the Brain CareNotes app or an attention control education-only app (Dementia Guide Expert) for 12 months.

The primary objective is to test the the usability and acceptability, as well as needs met and unmet by Brain CareNotes among Hispanic caregivers of persons with dementia. Barriers in access and acceptance of dementia care resources have been previously identified including gaps in understanding of beliefs or practices between patients and local health systems, low health literacy, language barriers, and other cultural factors. These barriers may affect usability and acceptance of interventions. Therefore, it is hypothesized that average scores on the Simplified Systems Usability Scale will be less than 70 and low acceptance rates will be reported by more than 70% of the Hispanic co-hort. These measures will be administered at 3, 6 and 12 months.

The secondary objective is to examine the needs of Hispanic caregivers that are met and unmet by the Brain CareNotes intervention. Information on how unique culturally influenced needs were met or not met by Brain CareNotes will be collected and suggestions for changes to the intervention app will be identified. This aim will be addressed qualitatively by providing semi-structured interviews guided by the PROGRESS-PLUS framework to the Hispanic participants who received the Brain CareNotes intervention (n=20) about their experience with the intervention and suggestions for changes. The PROGRESS-PLUS framework addresses cultural and socio-economic factors that should be considered when creating behavioral interventions that are culturally compatible. It is expected that responses to interviews will identify themes consistent with a lack of cultural compatibility to factors identified by the PROGRESS-PLUS framework.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* Self-identified primary unpaid Hispanic caregiver of a person diagnosed with ADRD (at any stage) who are:
* Receiving primary care and
* Community-dwelling;
* English literate;
* Age ≥ 18 years

Exclusion Criteria:

* Care recipient is a permanent resident of an extended care facility (nursing home);
* Involvement in another clinical trial that would prevent or interfere with study objectives;
* Sensory or other impairment prohibiting the use of a mobile touchscreen device or other study activity (after correction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | 3 months, 6 months,12 months
  10-item standardized survey of user-reported technology usability, based on revised System Usability Scale, with scale score computed ranging from 0-100, with 100 indicating highest possible perceived usability.
Behavioral Intention Questionnaire | 3 months, 6 months, 12 months
  A 4-item questionnaire assessing a user's intention to use a technology in the near future. Scores range from 0-24 with a high score representing greater intention to use the technology.

SECONDARY OUTCOMES:
Qualitative Interview | 12 months
  Participants in the intervention group will complete semi-structured interviews guided by the PROGRESS-PLUS framework. The purpose of these interviews will be to determine their needs that were met or not met by the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Holden, PhD, Principal Investigator — Indiana University; Malaz Boustani, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No